CLINICAL TRIAL: NCT05397457
Title: Effect of Helmet Type, Home-use Photobiomodulation Therapy Device for Chemotherapy-induced Alopecia
Brief Title: Effect of Helmet Type, Home-use Low-level Light Therapy Device for Chemotherapy-induced Alopecia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, YUAN-CHIEH YEH, Deputy Director, Assistant professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202200395A3
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Chemotherapy-induced Alopecia
MeSH Terms: conditions — Breast Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Device: low-level light therapy
- Control group (No Intervention)

INTERVENTIONS:
Device: low-level light therapy — Device: Hair Boom 69
  All participants within the experimental group will undergo low-level light therapy sessions 3 times a week for the total duration of 4 weeks starting at their last CT administration.
  If the participants can not cooperate to receive the therapy 3 times a week due to personal reasons, we will recommend that they undergo 2 courses of the therapy per week at least and finish the 12 courses of the intervention in 6 weeks.
  Arms: Treatment group

SUMMARY:
As far as breast cancer is concerned, chemotherapy (CT) is an important treatment. However, there are many adverse effects impairing the patient's quality of life (QOL), in which chemotherapy-induced alopecia (CIA) affects up to 65% of the patients. This condition is reversible. Nevertheless, it takes several months after CT for visible hair regrowth. Different characteristics of the new hair are common; for example, 65 percent of the patients have experienced a graying, curling, or straightening effect. Besides, the emotional trauma due to alopecia can not be neglected.

Currently, scalp cooling is the only available and verified management for prevention. Unfortunately, the success rate of scalp cooling is variable, especially among the patients receiving anthracycline-based combinations.

Low-level light therapy (LLLT) has been proven as a therapeutic technique for adrenergic alopecia. Recently, investigators have checked the validity of LLLT for the CIA. Although the preliminary outcome showed failure at accelerating hair recovery, technical progress of LLLT may improve the end result. Specifically, LLLT is a technique that utilizes laser diodes (LD) or light-emitting diodes (LED) to promote tissue repair. The light source from LD is coherent while LED is an incoherent light source. Therefore, LDs can deliver energy to tissues more efficiently than LEDs. To comprehensively evaluate the beneficial effect of LLLT in treating CIA, we conduct a clinical trial with a more advanced device equipped with 69 LDs.

The project aims to explore the effect of low-level light therapy in chemotherapy-induced alopecia. We expect the therapy will lead to an improvement in the patient's hair count, hair width, and quality of life after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 75 years
* Informed Consent as documented by signature.
* Able to read and converse in chinese
* Female
* Diagnosis of breast cancer
* They completed chemotherapy no more than 2 weeks
* Treatment with neoadjuvant (preoperative) or adjuvant (postoperative) chemotherapy: anthracycline and taxane containing (paclitaxel or docetaxel) chemotherapy regimen.
* life expectancy was at least 6 months.
* Diagnosed with CIA grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE)

Exclusion Criteria:

* scalp tumor or melanoma
* having any serious mental illness or history, or taking psychotropic drugs
* a medical history of dermatosis
* severe liver and kidney damage
* Pregnancy
* Take any of the following medications for 6 months prior to initiation of the study: topical minoxidil, and spironolactone, and topical calcitriol
* Receiving scalp cooling during chemotherapy

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 106 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hair counts recorded by Sentra scalp analyzer | Baseline
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair counts in the frontal, parietal, and occipital regions.
Hair counts recorded by Sentra scalp analyzer | 12th course of intervention (four weeks after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair counts in the frontal, parietal, and occipital regions.

SECONDARY OUTCOMES:
Chemotherapy-Induced Alopecia Distress Scale | Baseline
  A validated questionnaire was developed by the Korean Organization for Researching distress due to chemotherapy-induced alopecia.
  The minimum and maximum scores on the chemotherapy-induced alopecia distress scale are 17 and 68, respectively, including 17 items in 4 factors (Physical, emotional, activity, and relationship). The higher value suggests higher chemotherapy-induced distress that the participants encountered.
Chemotherapy-Induced Alopecia Distress Scale | 12th course of intervention (four weeks after the first course of intervention)
  A validated questionnaire was developed by the Korean Organization for Researching distress due to chemotherapy-induced alopecia.
  The minimum and maximum scores on the chemotherapy-induced alopecia distress scale are 17 and 68, respectively, including 17 items in 4 factors (Physical, emotional, activity, and relationship). The higher value suggests higher chemotherapy-induced distress that the participants encountered.
Rosenberg Self-esteem Scale | Baseline
  Self-esteem will be measured by Rosenberg's Self-Esteem scale with 10 items. Each item is scored on a 4-point Likert self-report scale, ranging from 0 to 3. A total score is obtained by summing all item scores. The minimum and maximum scores on the scale are 0 and 30. Scoring less than 15 may indicate problematic low self-esteem.
Rosenberg Self-esteem Scale | 12th course of intervention (four weeks after the first course of intervention)
  Self-esteem will be measured by Rosenberg's Self-Esteem scale with 10 items. Each item is scored on a 4-point Likert self-report scale, ranging from 0 to 3. A total score is obtained by summing all item scores. The minimum and maximum scores on the scale are 0 and 30. Scoring less than 15 may indicate problematic low self-esteem.
European Quality of Life 5 Dimensions 5 Level Version | Baseline
  The European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems, indicating his/her health state by ticking the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined into a 5-digit number describing the respondent's health state and divided into 5 levels of perceived problems:
  Level 1: no problem Level 2: slight problems Level 3: moderate problems Level 4: severe problems Level 5: extreme problems
European Quality of Life 5 Dimensions 5 Level Version | 12th course of intervention (four weeks after the first course of intervention)
  The European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems, indicating his/her health state by ticking the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined into a 5-digit number describing the respondent's health state and divided into 5 levels of perceived problems:
  Level 1: no problem Level 2: slight problems Level 3: moderate problems Level 4: severe problems Level 5: extreme problems
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | Baseline
  The European Organization for the Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  The 30-item questionnaire measuring QLQ (QLQ-C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. The high scale score represents a high response level.
  Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | 12th course of intervention (four weeks after the first course of intervention)
  The European Organization for the Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
  The 30-item questionnaire measuring QLQ (QLQ-C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. The high scale score represents a high response level.
  Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems
Hair width recorded by Sentra scalp analyzer | Baseline
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair width in the frontal, parietal, and occipital regions.
Hair counts recorded by Sentra scalp analyzer | 3rd course of intervention (one week after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair counts in the frontal, parietal, and occipital regions.
Hair width recorded by Sentra scalp analyzer | 3rd course of intervention (one week after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair width in the frontal, parietal, and occipital regions.
Hair counts recorded by Sentra scalp analyzer | 6th course of intervention (two weeks after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair counts in the frontal, parietal, and occipital regions.
Hair width recorded by Sentra scalp analyzer | 6th course of intervention (two weeks after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair width in the frontal, parietal, and occipital regions.
Hair counts recorded by Sentra scalp analyzer | 9th course of intervention (three weeks after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair counts in the frontal, parietal, and occipital regions.
Hair width recorded by Sentra scalp analyzer | 9th course of intervention (three weeks after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair width in the frontal, parietal, and occipital regions.
Hair width recorded by sentra scalp analyzer | 12th course of intervention (four weeks after the first course of intervention)
  Sentra scalp analyzer is an innovative phototrichogram, combining the technique of trichoscopy, image capture, and image interpretation. This device can be utilized to measure hair counts and hair width. We will record hair width in the frontal, parietal, and occipital regions.

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Derived] Wu CX, Li CH, Shiao YH, Cheng HY, Wu TH, Lee CH, Chang ZY, Yeh YC. The effect of a helmet type, home-use low-level light therapy device for chemotherapy-induced alopecia: study protocol for a randomized controlled trial. Trials. 2023 Dec 5;24(1):789. doi: 10.1186/s13063-023-07823-x. PMID 38053197